CLINICAL TRIAL: NCT01486888
Title: A Randomised, Single Centre, Double-blind, Two-period Cross-over, Glucose Clamp Trial to Test for Bioequivalence Between Insulin Mixtard® 30 (600 Nmol/ml) and Insulin Mixtard® 30 (1998 Nmol/ml) in Healthy Subjects
Brief Title: Bioequivalence of Two Mixtard® 30 Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX1000-1735; 2005-006050-24 (EudraCT Number)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — biphasic human insulin 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental)
  Interventions: Drug: biphasic human insulin 30
- Formulation B (Active Comparator)
  Interventions: Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic human insulin 30 — Single dose of each formulation, administered subcutaneously (s.c., under the skin) on two separate dosing visits

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to to test for bioequivalence between two formulations of Mixtard® 30 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2, inclusive
* Non-smoker, defined as no nicotine consumption for at least one year
* Fasting plasma glucose below or equal to 100 mg/dL (5.6 mmol/L)

Exclusion Criteria:

* Previous participation in this trial or other clinical trials within the last 3 months
* Body weight above 87.5 kg
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (intrauterine device (IUD) that has been in place for at least 3
* History of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin concentration-time curve (AUC 0-24 hours)
Maximum serum insulin concentration (Cmax)

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve (AUC 0-6 hours)
Area under the serum insulin concentration-time curve (AUC 6-24 hours)
Area under the serum insulin concentration-time curve (AUC 0-inifinity hours)
Time to maximum serum insulin concentration (tmax)
Terminal insulin half life (t½)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com